CLINICAL TRIAL: NCT06388122
Title: DiviTum®TKa: A Biomarker Assay for Efficacy in HR+ Metastatic Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-009689; NCI-2024-03405 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); MC240301 (Other: Mayo Clinic)
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: HER2-negative Breast Cancer; Hormone-receptor-positive Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1 (initiating 1st line CDK4/6 & endocrine therapy): Blood will be drawn every 14 days starting from the first treatment cycle until the start of cycle 3; starting at cycle 3 blood will be drawn the first day of every cycle thereafter until progression. Optional blood draws will be taken with standard of care labs when starting next therapy.
  Interventions: Procedure: Biospecimen Collection
- Group 2 (initiating 2nd or later line of CDK4/6 with or without endocrine therapy): Blood will be drawn every 14 days starting from the first treatment cycle until the start of cycle 3; starting at cycle 3 blood will be drawn the first day of every cycle thereafter until progression. Optional blood draws will be taken with standard of care labs when starting next therapy.
  Interventions: Procedure: Biospecimen Collection
- Group 3 (currently receiving 1st line CDK4/6 and endocrine therapy): Blood will be drawn on day 15 of the next cycle after enrollment and the first day of every cycle thereafter until progression. Optional blood draws will be taken with standard of care labs when starting next therapy.
  Interventions: Procedure: Biospecimen Collection
- Group 4 (initiating or currently receiving 1st or 2nd line endocrine therapy): Blood will be drawn at baseline or the first day of the treatment cycle and the first day of every cycle thereafter until progression. Optional blood draws will be taken with standard of care labs when starting next therapy.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
The purpose of this study is to explore the clinical utility of routinely measuring thymidine kinase activity (TKa) in HR+ metastatic breast cancer patients receiving treatment with any approved endocrine therapy either alone or in combination with any approved CDK4/6 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Pre- or post-menopausal HR+ metastatic breast cancer patients who are:

  * Group 1: scheduled to initiate 1st line combination therapy with an FDA-approved CDK4/6 inhibitor (palbociclib, ribociclib, or abemaciclib) and an FDA-approved endocrine therapy for pre- or post-menopausal HR+ metastatic breast cancer (mBC).
  * Group 2: scheduled to initiate second or later lines of therapy with an FDA-approved CDK4/6 inhibitor (palbociclib, ribociclib, or abemaciclib) with or without an FDA-approved endocrine therapy for pre- or post-menopausal HR+ mBC.
  * Group 3: currently receiving 1st line therapy with an FDA-approved CDK4/6 inhibitor (palbociclib, ribociclib, or abemaciclib) and an FDA-approved endocrine therapy for pre- or post-menopausal HR+ mBC.
  * Group 4: scheduled to initiate, or are currently receiving, 1st or 2nd line therapy of an FDA approved endocrine therapy (single agent) for pre- or post-menopausal HR+ mBC.

NOTE: Patients that meet eligibility criteria for any of the above groups that are already enrolled in an ongoing clinical trial are eligible for co-enrollment to this observational study.

Exclusion Criteria:

* Treatment including investigational agent or therapies
* Early breast cancer diagnosis
* Male breast cancer
* Currently receiving treatment for other active malignancy at time of registration

  * EXCEPTIONS: Nonmelanoma skin cancer or carcinoma-in-situ (e.g. of cervix, prostate)
* Inability to give written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients > 18 years old with diagnosis of metastatic HR positive HER2 negative breast cancer that will be or are currently being treated with standard of care endocrine therapy +/- CDK 4/6 inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2031-06-15 (Estimated); Study Completion 2031-06-15 (Estimated)

PRIMARY OUTCOMES:
DiviTum®TKa assay as an early predictor of primary treatment resistance | Every cycle (approximately 28 days) until disease progression up to 6 months
  Blood samples collected from participants will be assessed using DiviTum®TKa assay for thymidine kinase activity (TKa) levels above Limit of Detection (LOD) as a predictor of primary treatment resistance. Primary treatment resistance will be defined as disease progression in less than 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Advani, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials